CLINICAL TRIAL: NCT05512559
Title: Value of Body Composition Analysis in Predicting Delayed Emergence From Remimazolam-based General Anesthesia: A Prospective Observational Study.
Brief Title: Body Composition Analysis and Time to Emergence From Remimazolam
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hwan Lee, Professor, Samsung Medical Center
Other Study IDs: SMC 2022-06-074
Record Dates: First submitted 2022-08-21; First posted 2022-08-23 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Remimazolam; Body Composition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- remimazolam: general anesthesia induction with 6mg/kg/hr continuous infusion of remimazolam. general anesthesia maintenance with 1mg/kg/hr continuous infusion of remimazolam.
  Interventions: Device: body composition analysis

INTERVENTIONS:
Device: body composition analysis — Body composition analysis by bioelectrical impedance measurement, just before induction of anesthesia.

SUMMARY:
Remimazolam is a novel general anesthetic drug. The time to emergence from remimazolam-based general anesthesia is variable among patients, but little is known about the risk factors for delayed emergence. We believe that information from body composition analysis may be helpful in understanding which patients are more likely to show delayed emergence from remimazolam.

ELIGIBILITY:
Inclusion Criteria:

* Adult ASA I-III patients undergoing cerebral aneurysm coil embolization under general anesthesia using remimazolam

Exclusion Criteria:

* Patients with preoperative mental change, hemodynamic instability, hemodialysis, heart failure, hypoalbuminemia, pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ASA I-III patients undergoing cerebral aneurysm coil embolization under general anesthesia using remimazolam
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
emergence time | at the time of emergence
  relationship between body composition analysis information and time to emergence after discontinuing remimazolam infusion.

SECONDARY OUTCOMES:
time to loss of consciousness | at the time of induction
  relationship between body composition analysis information and time to loss of consciousness after starting remimazolam infusion.
hypotension | from induction to emergence of anesthesia
  relationship between body composition analysis information and hypotensive event during anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Sungkyunkwan University, School of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided